CLINICAL TRIAL: NCT04355481
Title: Study of the Dissemination of SARS-COV-2 in the Environment of Infected Patients Admitted to Intensive Care Unit
Brief Title: Dissemination of SARS-COV-2 (COVID-19) in the Environment of Infected Patients Admitted to Intensive Care Unit
Acronym: ENVIROREA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200411; 2020-A00897-32 (Registry Identifier: ANSM IDRCB number)
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Covid-19; Viral Infection
Keywords: SARS-Cov-2; environmental contamination; intensive care unit
MeSH Terms: conditions — COVID-19; Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this protocol is to estimate the proportion of patients hospitalized in intensive care unit for a SARS-Cov-2 viral lung infection and contaminating their environment at 1 meter. The contamination will be assessed by quantifying the viral RNA by RT-PCR on a 600-liter air sample aspirated by a Coriolis® system. This sample will be taken within 48 hours after the confirmation of SARS-Cov-2 infection, documented by RT-PCR. In fact, the hospital hygiene measures practiced in intensive care unit in patients with viral respiratory infection are identical to those practiced in other services. These measures are possibly insufficient as evidenced by recent data related to the COVID-19 epidemic.

DETAILED DESCRIPTION:
Respiratory viruses are frequently responsible for acute respiratory failure which justifies hospitalization in intensive care unit. Actually, recent epidemics of emerging viruses (including COVID-19) have highlighted the possibility of air-type transmission in this specific population. Despite the fact that the risk of environmental contamination has never been objectified, It is probable that in intensive care patients, this contamination is greater than in other patients because of the gravity of the patients (greater inoculum) and the use of ventilation techniques responsible for probably increased exhaled viral expression. Defining the mode of transmission of respiratory viruses has major consequences in terms means of prevention. The "air" mode of transmission absolutely requires hospitalization in a single room and sometimes additional air treatment. The droplet transmission mode due to its short range requires simpler measures (wearing a surgical mask, no specific air treatment) and has also led to the discussion of the value of the individual room. Indeed, the use of high flow ventilation system such as "optiflow" or non-invasive ventilation, can transform a droplet risk into "air" risk. For this reason, measuring the extent of environmental contamination around infected patients in intensive care is a major issue.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old.
* Patient admitted to intensive care unit for a low respiratory infection during which the SARS-Cov-2 virus is documented, with a positive RT-PCR in the 48 hours before taking samples.
* Information and not opposition from the patient / or family

Exclusion Criteria:

* No documentation of SARS-Cov-2 viral respiratory infection.
* Patient under guardianship / curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are recruited at the intensive care unit, for all patients admitted to intensive care for a low respiratory infection during which the SARS-Cov-2 virus (RT-PCR positive) is documented within 48 hours before carrying out the air and surfaces specimens.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-04-17 (Actual); Primary Completion 2020-10-17 (Estimated); Study Completion 2020-12-17 (Estimated)

PRIMARY OUTCOMES:
Estimate the proportion of patients hospitalized in intensive care for a SARS-Cov-2 viral lung infection and contaminating their environment at 1 meter. | within 48 hours of the confirmation of SARS-Cov-2 infection documented by RT-PCR
  The primary objective of the study will be evaluated by the proportion of patients contaminating the air 1 meter from their face.
  The contamination will be assessed by quantifying the viral RNA by RT-PCR on a 600-liter air sample aspirated by a Coriolis® system. This sample will be taken within 48 hours after the confirmation of SARS-Cov-2 infection, documented by RT-PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Yacine TANDJAOUI-LAMBIOTTE, Dr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (3):
- France (3):
  - Service de réanimation Hôpital Avicenne, Bobigny
  - Service de réanimation Hôpital Bichat, Paris
  - Service de réanimation Hôpital Tenon, Paris